CLINICAL TRIAL: NCT04857944
Title: Personalised Exercise Prescription: the Efficiency of a Transdisciplinary Blended Intervention in Depressive Symptoms
Brief Title: Improving Depressive Symptoms Through Personalised Exercise and Activation
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar Research Institute (IMIM) (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Francesc Colom, Group leader and senior researcher, Hospital del Mar Research Institute (IMIM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI19/00009
Record Dates: First submitted 2021-04-16; First posted 2021-04-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Depressive Symptoms; Depressive Disorder
Keywords: Depressive symptoms; Exercise; Personalized medicine; Blended intervention; Transdisciplinary
MeSH Terms: conditions — Depression; Depressive Disorder; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After assignment to study conditions, participants and investigators will be blinded to one aspect of the specific experimental intervention (receiving or not motivational messages). Both will know whether participants have been allocated to experimental or control conditions but the specific experimental intervention (A or B) will not be revealed. To avoid assessment bias, an independent evaluator blinded to group allocation will complete follow-up assessments.
  Clinicians, principal investigators, and statisticians will be also blinded to the randomization procedure and group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalised exercise group program + fitness tracker + app with motivational messages (A) (Experimental): After study entry and baseline assessments, subjects will attend the one-month IDEA group sessions aimed at promoting physical activity and exercise. Participants randomly assigned to this study arm will use the smart band and the app with the motivation set enabled, allowing participants to receive the messages according to their compliance and adherence to the personalised prescriptions. After group sessions (week 4), study subjects will start receiving motivational messages up until the end of the trial (8 consecutive months).
  Interventions: Behavioral: IDEA program (Improving depressive symptoms through personalised exercise and activation); Device: IDEApp
- Personalised exercise group program + fitness tracker + app without motivational messages (B) (Experimental): Subjects will follow the same procedure as intervention A, with the difference that the app will have the motivation set disabled, therefore participants will not receive any messages regarding their compliance. After group sessions, study subjects will be expected to continue using the smart band and app up until the end of the trial (8 consecutive months).
  Interventions: Behavioral: IDEA program (Improving depressive symptoms through personalised exercise and activation); Device: IDEApp
- Fitness tracker + app without motivational messages (CG) (Sham Comparator): After study entry and baseline assessments, all patients assigned to the control group will receive both the app and the smart band, but the motivation set will be disabled. Study subjects will be expected to use the smart band and app up until the end of the trial.
  Interventions: Device: IDEApp

INTERVENTIONS:
Behavioral: IDEA program (Improving depressive symptoms through personalised exercise and activation) — The program will consist of six 90-minute group sessions composed of four to six participants. These short intervention sessions will be distributed in one month, with a frequency of once or twice a week depending on the week of the program. Of the six sessions, two will be exercise-oriented and will include on-site practice. The remaining four sessions will include definitions of depressive symptomatology, the relationship between depression and having an active lifestyle, motivation and barriers towards exercise, and maintenance strategies.
  Arms: Personalised exercise group program + fitness tracker + app with motivational messages (A); Personalised exercise group program + fitness tracker + app without motivational messages (B)
Device: IDEApp — An ad-hoc app (IDEApp) combined with a fitness tracker to register and store participants' physical activity, exercise compliance, and sleep patterns. The app will deliver motivational or awareness messages when the fitness tracker detects non-compliance with the exercise prescription, physical activity decreases, or altered sleep patterns.

SUMMARY:
The purpose of the present study is to evaluate the changes on mental and physical health deriving from a blended intervention merging psychological intervention aimed at increasing activity and exercise with a personalised exercise program based on medical assessment on subjects suffering from mild to moderate depressive symptoms irrespective of diagnostic entity, by comparing two experimental groups (A. Personalised exercise group program+ app with motivational messages + fitness tracker or B. Personalised exercise group program+ app with no motivational messages + fitness tracker) and a control group (app with no motivational messages +fitness tracker). This study also introduces the use of a wearable device to collect information regarding physical activity and sleep patterns to provide motivational messages.

The investigators hypothesise that participation in a brief app-blended group intervention -on top of usual care- promoting personalised exercise and activity will improve functioning and well-being of participants, as well as motivate them to increase their physical activity and enhance behavioural changes towards a healthier lifestyle when compared to general exercise prescriptions. In addition, the investigators hypothesise that amongst patients who had been allocated to the intervention conditions, those presenting better commitment to prescribed personalised exercise plans (understood as more than a 70% compliance of prescribed exercise, measured by objective movement data collected by a fitness tracker) will show a higher functionality improvement.

DETAILED DESCRIPTION:
OBJECTIVE

Primary:

·To evaluate the changes on functioning deriving from a blended intervention merging psychological intervention aimed at increasing activity and exercise with a personalised exercise program based on medical assessment on subjects suffering from mild to moderate depressive symptoms.

Secondary:

* To test the differential effect of the above-mentioned blended exercise program on wellbeing, depressive symptoms and physical activity performance of patients with depressive symptoms, by comparing the three study arms.
* To measure wellbeing of patients allocated to the personalised exercise program, compared to the group condition.
* To assess and compare antidepressive response within both groups and intra subject at interim visits and final assessment.
* To measure effects of a personalised exercise program on exercise capacity and strength.

Exploratory:

· To study gender differences concerning all treatment outcome parameters.

STUDY DESIGN The investigators will conduct a 3-arm randomized controlled clinical trial in which eligible participants will be allocated to one of the following conditions: a)Intervention A: Personalised exercise group program + fitness tracker + IDEApp with motivational messages; b)Intervention B: Personalised exercise group program + fitness tracker + IDEApp without motivational messages; c) Control Group: fitness tracker +IDEApp without motivational messages.

All participants, regardless of their treatment condition, will be read a short text about the the benefits of regular exercise on mood during the initial clinical interview, in order to make sure that they have listened to this unspecific advice at least once.

This study seeks to investigate the effects of personalised exercise on top of usual care. All participants will continue receiving naturalistic pharmacological and/or psychological treatment, without any research-related disruption.

TARGET POPULATION Male and female patients with current depressive symptoms regardless of diagnosis entity.

SETTING Outpatient mental health centres and General Practice(GP) surgeries belonging to the healthcare network of Hospital del Mar in Barcelona, Spain. Referrals will be made by any general practitioner, nurse, psychologist or psychiatrist treating the patient. Group sessions will be facilitated by a psychologist (Psychology BSc, MSc) and a physiotherapist (Physiotherapy BSc, MSc) who will undertake brief and intuitive therapy training.

Before any study procedures occur, participants will be informed about the study characteristics, will be provided with a study information leaflet and a written informed consent form must be signed by them. After signing the informed consent, a competent practitioner will confirm or disregard depressive symptomatology, administer the MADRS and judge that the subjects fulfil all the inclusion criteria items and none of the exclusion criteria requirements.

INTERVENTION The main goal of the intervention is to personalise exercise prescription and enhance motivation towards being physically active. To fulfil our objectives, a collaborative team of psychologists, Physical Medicine and Rehabilitation specialists, and one psychiatrist developed a brief group intervention -the IDEA programme- and an ad-hoc made app to register and store the participants' physical activity, exercise compliance and sleep patterns.

In the exercise-oriented sessions, participants will be asked to wear sports clothes to practice the individualised exercise prescription on-site and will receive an individual brochure with indications and photographs of their prescription.

For the implementation of the sessions, the research team developed a guide for the professionals with the content of each session and its dynamics. In the case of the individualised exercise prescription, a pool of exercises was created in order to standardize the potential exercises that will be chosen individually for each participant.

MOBILE APPLICATION DEVELOPMENT A collaborative team of psychologists, Physical Medicine and Rehabilitation specialists and software engineers developed a user-friendly smartphone application (IDEApp) that can be synchronised to a fitness tracker. The fitness tracker will register and store data regarding physical activity and sleep patterns. IDEApp will collect two types of data: objective and self-informed. Objective data will include the number of daily steps, aerobic exercise -including minutes, distance in metres, maximum, minimum and average heart rate- and sleep structure -including duration in a 24-hour period, deep and light sleep discrimination-. Self-reported data will require participants to simply indicate on IDEApp whether one of three exercise options have been performed: 1) relaxation, 2) stretching, or 3) strength and endurance.

When non-compliance with the exercise prescription, physical activity decreases, or altered sleep patterns are detected, the system will trigger motivational or awareness messages through the app.

NUMBER OF SUBJECTS 172 participants with mild to moderate depressive symptoms irrespective of diagnosis entity will complete the study.

RECRUITMENT The recruitment period will extend over 12 months and all participants will be given away an activity band that will be free to use together with free access to the app after study completion.

IMPLEMENTATION Allocation and intervention assignment will be automatically generated by the IDEApp web-based platform once participants are registered in the system by study staff. Participants will be enrolled in the trial by a study psychologist after baseline assessment.

ASSESSMENT Participants will attend the study entry clinical interview and baseline assessment, followed by an evaluation with a physiotherapist to identify their physical needs and capabilities. Such assessments will allow the subsequent prescription of tailored exercise to the intervention groups. After baseline assessment, the study staff will install IDEApp on the smartphone of all participants and provide them with the activity band. In the first week after study entry, all subjects will effectively start using the devices and IDEApp, which will provide estimates of their baseline physical activity and exercise, and up until the end of the trial.

After group sessions completion (after 1 month for Control Group), every participant will be followed by an eight-month follow-up. Post-allocation assessments following the intervention at 4-weeks (T1) and 12-weeks (T2) will be carried out by telephone. The final assessment at 36-weeks (T3) will be carried out face-to-face and will follow a similar outline as the baseline assessment.

DATA MANAGEMENT Study data will be collected, entered and managed using REDCap electronic data capture tools hosted at Hospital del Mar Medical Research Institute (IMIM). More specifically, data will be collected offline in the REDCap mobile app on an Android tablet and then will be sync back to the project on the REDCap server. A password system will be utilized to control access to data and the activity that researchers may undertake is regulated by the privileges associated with their user identification code.

STATISTICAL ANALYSIS PLAN FOR PRIMARY AND SECONDARY OUTCOMES Statistical analysis will be performed using the software SPSS Statistics 25. Descriptive statistics will be used to analyse the distribution of socio-demographic and clinical characteristics among groups at baseline. Continuous variables with a normal distribution will be analysed performing an ANOVA. Where the premises of normalcy are not met, the Wilcoxon test will be used. The differences between groups on the categorical and mail clinical variables will be evaluated by using a Chi-square test. Those variables that are statistically significant may be used as covariates for a logistic or linear regression study of the factors associated with the magnitude of the effect, and determine which variables are better predictors of functioning. The effect size index will be estimated in case of correlation indexes for each of the performed analyses. To analyse efficacy the investigators will perform intention to treat analysis. Analysis will be two-tailed and the significance set a p <0.05.

Last Observation Carried Forward analysis will be used to handle and minimize missing data on the clinical variables.

ENDPOINTS

Primary endpoint

●Change in psychosocial and occupational functioning of subjects allocated to both the experimental conditions (A+B) versus control condition, as measured by the SF-36 from baseline to week 36 and from baseline to interim visits.

Secondary endpoints

* Improvement in wellbeing of subjects allocated to both the experimental conditions (A+B), as measured by the WHO-5 Well-Being Index (WHO 5 WBI) from baseline to week 36 and from baseline to interim visits.
* Improvement in depressive symptoms of subjects allocated to both the experimental conditions (A+B), as measured by the Patient Health Questionnaire (PHQ-9) from baseline to week 36 and from baseline to interim visits.
* Improvement in current physical activity of subjects allocated to both the experimental conditions (A+B), as measured by the Simple Physical Activity Questionnaire (SIMPAQ) from baseline to week 36 and from baseline to interim visits.
* Change in functional exercise capacity using the 6-minutes walking test (6MWT) from baseline to week 36 in subjects receiving experimental conditions (A+B) of personalised exercise prescription versus control condition. The change in the distance walked in the 6MWT after completion of the program will be used to evaluate the effectiveness of the personalised exercise program. For the evaluation of dyspnea and subjective fatigue, the short Borg CR 10 Scale will be used before and after the test.
* Change in functional exercise capacity using the 1-min STS test from baseline to week 36 in subjects receiving experimental conditions (A+B) of personalised exercise prescription versus control condition.
* Change in isometric muscle strength of the hand and the forearm using the handgrip strength test from baseline to week 36 in subjects receiving experimental conditions (A+B)of personalised exercise prescription versus control condition. The equipment used will be a Jamar Plus+ digital hand dynamometer, grip strength will be measured 3 times per hand in the 2-handle position.
* Proportion of participants allocated to the experimental conditions (A+B) presenting better commitment to prescribed personalised exercise plans -understood as more than a 70% compliance of prescribed exercise-measured by objective activity data recorded by the smartband-at follow-up visits.
* Change in physical activity and enhancement of a healthier lifestyle-as measured by activity and sleep objective data provided by a smartband and an ad-hoc-designed app- from baseline to week 36.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18-<65 years
* Presenting mild to moderate depressive symptoms according to Montgomery-Asberg Depression Rating Scale (MADRS score>16 & <34)
* Currently owning an Android compatible smartphone
* Fluent in the Spanish language
* Basic knowledge and skills using information and communication technology
* Be able to provide written informed consent to participate

Exclusion Criteria:

* Severe cognitive and/or physical impairment
* Cognitive deficit or developmental disorder
* Current psychotic, melancholic, or catatonic features
* Drug or alcohol abuse
* Modification of drug treatment (or its dose) in the last month (or plan for it
* Beginning of psychological treatment in the last month
* Beginning of biophysical treatment in the last month
* BMI >40
* Physical disability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Psychosocial and occupational functioning | Baseline, 4 weeks, 12 weeks, and 36 weeks.
  The Functioning Assessment Short Test (FAST) will be used to assess the change in psychosocial and occupational functioning comparing subjects allocated to both experimental conditions (A+B) vs the control condition.
  The FAST is a simple self-administered instrument that comprises 24 items. It assesses impairment or disability in six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time.

SECONDARY OUTCOMES:
Depressive symptomatology | Baseline, 4 weeks, 12 weeks, and 36 weeks.
  The Patient Health Questionnaire (PHQ-9) will be used to assess the severity and improvement of depressive symptomatology.
  The PHQ-9 is a self-administered questionnaire used to screen the presence and severity of depression. It has 9 items on a scale from 0 (not at all) to 3 (nearly every day), the total score ranges from 0 to 27, with higher scores meaning severe depressive symptomatology.
Well-being | Baseline, 4 weeks, 12 weeks, and 36 weeks.
  Well-being will be assessed by the World Health Organization Well-Being Index (WHO-5).
  The WHO-5 a 5-item self-administered questionnaire used to assess current mental well-being. The rating scores go from 0 (at no time) to 5 (all of the time), with total scores ranging from 0 to 100, where higher scores mean the best imaginable well-being.
Exercise motives | Baseline to week 36.
  The Exercise Motivations Inventory (EMI-2) will be used to identify participants' motives to initiate and adhere to the personalised exercise prescription, and if they have changed during the trial.
  The EMI-2 is a 51-item, self-administered questionnaire used to assess the motives that are related to the practice of exercise. The rating scores go from 0 (not true at all for me) to 10 (totally true for me). Scores can be interpreted according to three different options: analysing individual items, analysing the 5 main areas (psychological, interpersonal, health, appearance and physical form), or a global score. Higher scores on either option mean that those reasons are what motivate exercise practise.
Physical and social functioning | Baseline, 4 weeks, 12 weeks, and 36 weeks.
  The 36-item Short-Form Health Survey (SF-36) will be used to assess the change in physical and social functioning comparing subjects allocated to both experimental conditions (A+B) vs the control condition.
  The SF-36 is a 36-item, self-administered questionnaire used to assess general health status, and it includes eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The scores of each domain depend on the number of items in them; however, these scores are transformed on a scale from 0 to 100, where higher scores indicate less disability and better general health status.

OTHER OUTCOMES:
Physical Activity | Baseline, 4 weeks,12 weeks, and 36 weeks.
  The Simple Physical Activity Questionnaire (SIMPAQ) will be used to assess change in the percentage of practise of physical activity and sedentary time.
  The SIMPAQ is a 5-item clinical interview used to assess physical activity in a population at risk of high sedentary behaviour. The items assess time in bed, sedentary time, time spent walking, structured exercise and incidental or non-structured physical activity. It does not include scoring indications but aims to evaluate the physical activity to be able to increase it and reduce sedentary behaviour.
Aerobic capacity and endurance | Baseline to week 36.
  Changes in performance capacity assessed by the 6-Minutes Walking Test (6MWT). The 6MWT consists of measuring the distance a person can walk in the time frame of 6 minutes. There is no scoring instruction, as the results depend on individual variables and the own subject becomes its control.
  Heath rate, oxygen saturation, dyspnoea will be assessed before and after the test.
  To assess the fatigued cause by the test a reduced Borg scale will be used.
Functional exercise capacity and leg muscle strength | Baseline to week 36.
  Changes in exercise capacity and leg muscle strength evaluated by the 1-Min Sit to Stand Test (1MSTS).
  The 1MSTS consists of getting up from and sitting on a chair as fast as possible within one minute. The scoring includes counting how many times the person repeats the action. Fatigue perceived after the test will be rated using a modified Borg scale.
Functional exercise capacity and isometric muscle strength | Baseline to week 36.
  Changes in functional exercise capacity and isometric muscle strength will be assessed by the Handgrip Strength Test.
  The Handgrip Strength Test will be performed using a Jamar Plus+ digital hand dynamometer; grip strength will be measured three times per hand in the 2-handle position. A mean score of the three tries will be calculated, and the fatigue caused by the test will be assessed with the reduced Borg scale.
Activity and sleep patterns | Baseline to week 36.
  Changes in Activity and sleep patterns based on objective data collected by a fitness tracker (Xiaomi Mi Band 5). This wearable device will collect data including the number of daily steps, aerobic exercise (minutes, distance in meters, maximum, minimum, and average heart rate) and sleep structure (time of sleep per 24-hour period, deep and light sleep discrimination).

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duarte, Dr, Principal Investigator — Parc de Salut Mar; Francesc Colom, Dr, Principal Investigator — Parc de Salut Mar
Locations (1):
- Centre Fòrum (Consorci Mar Parc de Salut de Barcelona), Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Garcia-Estela A, Angarita-Osorio N, Alonso S, Polo M, Roldan-Berengue M, Messaggi-Sartor M, Mur-Mila E, Vargas-Puertolas L, Perez V, Duarte E, Colom F. Improving Depressive Symptoms through Personalised Exercise and Activation (IDEA): Study Protocol for a Randomised Controlled Trial. Int J Environ Res Public Health. 2021 Jun 10;18(12):6306. doi: 10.3390/ijerph18126306. PMID 34200805